CLINICAL TRIAL: NCT03377569
Title: Understanding the Role of Subcortical Oscillations in Human Sleep Dysregulation.
Brief Title: Subcortical Oscillations in Human Sleep Dysregulation
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 17-0868
Record Dates: First submitted 2017-11-29; First posted 2017-12-19 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease; REM Behavior Disorder
Keywords: Deep Brain Stimulation; Polysomnography; Actigraphy
MeSH Terms: conditions — Parkinson Disease; REM Sleep Behavior Disorder | interventions — Sleep

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group #1: Patients with Parkinsons Disease who will undergo Deep Brain Stimulation surgery. At home sleep monitoring prior to DBS surgery and in patient polysomnography with neural recording after DBS surgery.
  Interventions: Other: Sleep, PD and DBS
- Group #2: Patients with Parkinsons Disease who will undergo Deep Brain Stimulation surgery. At home sleep monitoring after DBS surgery with DBS stimulation on at night, and in patient polysomnography after DBS surgery.
  Interventions: Other: Sleep, PD and DBS
- Group #3: Patients with Parkinsons Disease who will undergo Deep Brain Stimulation surgery. At home sleep monitoring after DBS surgery with DBS stimulation off at night, and in patient polysomnography after DBS surgery.
  Interventions: Other: Sleep, PD and DBS

INTERVENTIONS:
Other: Sleep, PD and DBS — Sleep, PD and DBS

SUMMARY:
Sleep problems are common in the United States (US) adult population (>50 million), and have a negative impact on quality of life, productivity, and healthcare. A major obstacle to understanding how the brain is involved in human sleep disorders has been the lack of recordings of human brain function, from inside the brain, during the known sleep states.

DETAILED DESCRIPTION:
Sleep is necessary for life; critically important to the regulation of body and brain function. Sleep problems are common in the U.S. adult population (>50 million), and have a negative impact on quality of life, productivity, and healthcare. A major obstacle to understanding how the brain is involved in human sleep disorders has been the lack of recordings of brain function, from inside the brain, during the known sleep states; non-rapid eye movement (NREM) and rapid eye movement (REM). It is very common for patients with Parkinson's disease (PD) to also have sleep disorders, such as insomnia, restless-leg-syndrome and REM-behavior disorder. One treatment for PD patients is deep brain stimulation (DBS) of the subthalamic nucleus (STN-DBS). Despite evidence showing that STN-DBS improves several aspects of sleep behavior in PD subjects, few studies have examined the relationship between brain activity and sleep regulation in human subjects. In this proposal, the investigators will examine sleep in humans by recording brain activity from STN of PD patients who have undergone DBS surgery. The investigators will also test the hypothesis that STN contributes to both the regulation and disruption of normal sleep behavior.

ELIGIBILITY:
Inclusion Criteria:

Subjects with Parkinson's Disease (PD) who are planning to have staged, bilateral deep brain stimulation surgery at the University of Colorado Hospital and willing and able to do the following:

1. Have a computer and be willing to use it as part of this study.
2. Be able to learn to use and maintain a wristband-style sleep monitor.
3. Turn off their Implantable Pulse Generator (IPG, implanted battery).
4. Wear a wristband-style sleep monitor for 3 weeks, 6 weeks prior to surgery.
5. Spend one overnight research stay in the UCH Sleep lab, 3 weeks prior to DBS surgery .
6. Spend one overnight research stay in the UCH Sleep lab, immediately prior to IPG surgery, to record brain activity from the DBS electrode .
7. Have a 15 minute surgery to externalize the DBS lead cable to allow overnight recordings to occur.
8. Be pseudo-randomized to one of 2 conditions: OFF stimulation or ON stimulation.
9. Wear a wristband-style sleep monitor for 3 weeks, 3 months post-DBS surgery, in one of the 2 pseudo-randomized conditions.
10. Spend one overnight research stay in the UCH Sleep lab, 4 months post DBS surgery, in one of the pseudo-randomized conditions.

Subjects will have a sleep disorder documented in their medical history as determined by a single question screen for REM sleep behavior disorder.

Exclusion Criteria:

1. Subjects with Parkinson's Disease (PD) who are not planning to have staged, bilateral deep brain stimulation surgery at the University of Colorado Hospital.
2. Subjects without a documented sleep disorder.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinsons Disease and a documented sleep disorder planning on undergoing bilateral Deep Brain Stimulation surgery at the University of Colorado Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2020-08-02 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Measuring brain physiological activity via local field potentials and correlation to sleep states (REM, non-REM, etc.) | One entire sleep cycle (each cycle is 8-10 hours).
  STN LFP activity will be measured by externalized DBS electrodes during in patient polysomnography.
Chronic actigraphy to characterize sleep-wake behavior | 3 weeks
  The investigators will collect typical sleep-wake behavior-including indirect features of sleep disturbance-by equipping patients with a sleep-monitoring device (ActiGraph AW2) that will record sleep parameters.
Test the functional impact of STN-DBS on sleep-wake behavior through actigraphy | 3 weeks
  The investigators will examine the impact of STN modulation, via DBS in both On- and Off-Stimulation conditions in separate groups of subjects, on typical sleep-wake behavior.

CONTACTS AND LOCATIONS:
Overall Officials: John A Thompson, Ph.D., Principal Investigator — Principal Investigator
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No